CLINICAL TRIAL: NCT07161011
Title: Phase 2b, Proof-of-Concept, Single-center, Double-Masked, Randomized Study Comparing the Safety, Tolerability, and Efficacy of Three Different Ophthalmic Eyelid Wipe Dosing Techniques Using IVW-1001 in Subjects With Dry Eye Disease
Brief Title: Phase 2b Controlled Study of Dosing Techniques - Part B
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IVIEW Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVW-1001-CS-202B
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Dry Eye
Keywords: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Double-masked, randomized, parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IVW-1001 0.2% (Experimental): Ophthalmic Eyelid wipe
  Interventions: Drug: IVW-1001 Ophthalmic Eyelid Wipe 0.2%
- IVW-1001 0.4% (Experimental): Ophthalmic Eyelid Wipe
  Interventions: Drug: IVW-1001 Ophthalmic Eyelid Wipe 0.4%

INTERVENTIONS:
Drug: IVW-1001 Ophthalmic Eyelid Wipe 0.2% — Low dose
  Arms: IVW-1001 0.2%
Drug: IVW-1001 Ophthalmic Eyelid Wipe 0.4% — High dose
  Arms: IVW-1001 0.4%

SUMMARY:
Double-masked, dose-response of two concentrations of IVW-1001

DETAILED DESCRIPTION:
Using the best dosing technique from Study NCT07140380, subjects will be randomized to one of two concentrations.

ELIGIBILITY:
Inclusion:

Self-reported diagnosis of DED in one or both eyes

* BCVA +0.70 logarithm of minimum angle of refraction (Snellen equivalent 20/100) or better in each eye at the Screening Visit
* For women of childbearing potential, confirmed negative pregnancy test at the Screening Visit, not nursing a child, and willing to comply with one of the acceptable methods of birth control described in the protocol
* History (by subject recollection) of artificial tear use within 30 days prior to the Screening Visit
* Unanesthetized Schirmer's test score 5-19 mm inclusive in at least 1 eye (same eye) at the Screening Visit and the Baseline Visit

Exclusion Criteria:

* Corneal fluorescein staining score of 4 in either eye in any zone using the National Eye Institute grading system at either the Screening Visit or the Baseline Visit
* IOP ≥23 mmHg in either eye at either the Screening Visit or the Baseline Visit
* History of glaucoma or ocular hypertension in either eye requiring past or current medical or surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Unanesthetized Schirmer test | 7 days
  Tear production

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Research Foundation, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No